CLINICAL TRIAL: NCT06887569
Title: Using Financial Incentives and Screening to Increase Engagement With Mental Health Services Among College Students in Chennai, India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Harvard University (Other); University of California, Berkeley (Other); University of Michigan (Other); Institute for Financial Management and Research (Other); Abdul Latif Jameel Poverty Action Lab (Other); Schizophrenia Research Foundation (SCARF India), Chennai, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2206000666
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Depression/Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Information about mental health and therapy and free access to therapy
- Screening (Experimental): Information about screening for depression and anxiety. Information about mental health and therapy and free access to therapy
  Interventions: Behavioral: Screening
- Rewards (Experimental): Financial rewards for attending therapy. Information about mental health and therapy and free access to therapy
  Interventions: Behavioral: Rewards
- Screening + Rewards (Experimental): Information about screening for depression and anxiety, and financial rewards for attending therapy (combination of previous two treatments). Information about mental health and therapy and free access to therapy
  Interventions: Behavioral: Rewards; Behavioral: Screening

INTERVENTIONS:
Behavioral: Rewards — Financial rewards for attending therapy
  Arms: Rewards; Screening + Rewards
Behavioral: Screening — Information about screening for depression and anxiety
  Arms: Screening; Screening + Rewards

SUMMARY:
This study will evaluate the effectiveness of interventions to increase engagement with mental health services among a sample of college students in Chennai, India. The study is being conducted in partnership with an arts and science college for women in Chennai. The sample will be recruited within classrooms, during college hours. All students present in the classroom per the allotted time will be introduced to the study. The research team will obtain consent from those interested after screening them for age eligibility (between the ages of 18 and 30 years). Study participants will then complete a baseline survey including questions around demographics, perceptions of their own mental health, mental health treatment history, and the PHQ-ADS, a standardized composite screening tool for depression and anxiety. The experimental design is an RCT with 4 groups, randomized at the individual level: (1) a control group, which will watch a video with information about mental health and be able to access therapy in college and at SCARF, a mental health center in Chennai, at no cost for the duration of the study; (2) a screening group, in which, in addition to the interventions in the control group, students will be informed whether their responses to the PHQ-ADS questions fit in the standard risk categories of no, mild, moderate, or severe distress and corresponding recommendations for whether to make an appointment with a counselor/therapist; (3) a rewards group, in which, in addition to the interventions in the control group, students will be provided with a cash payment for attending their first therapy session; and (4) a combined screening and rewards group. The investigators will measure interest in, and take-up of, therapy at the individual level.

ELIGIBILITY:
Inclusion criteria:

* aged 18-30
* are present in the classrooms,
* consent to participate in the study

Exclusion criteria: None

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Proportion of participants expressing interest in therapy | Immediately after treatment (Day 1)
  Student stating interest in the participant survey in booking an appointment with a study counselor, or asking to be contacted by a study counselor to discuss mental health and therapy
Proportion of participants making an appointment | From enrolment until two months after enrolment
  student completing the process to make an appointment for therapy with a study counselor, through the participant survey or otherwise

SECONDARY OUTCOMES:
Proportion of participants taking-up of a mental health care app | Immediately after treatment (Day 1)
  This is measured in two ways: participants expressing interest in accessing a mental-healthcare app in the survey, and participants actually clicking a link to download the app.
Proportion of participants demanding for information about mental health | Immediately after treatment (Day 1)
  This is measured in two ways: participants expressing interest in receiving more information about mental health, and participants actually clicking a link to access the information
Proportion of participants attending therapy sessions | From enrolment until two months after enrolment
  Data will be collected from the administrative records of the counselling office on whether participants actually attended a therapy session, as well as the number of sessions attended.

OTHER OUTCOMES:
Proportion of participants reporting they would consider seeking therapy in future | Immediately after treatment (Day 1)
  Participants are asked whether they would consider seeking therapy in future
Proportion of participants reporting specific steps they would take to take care of their mental health | Immediately after treatment (Day 1)
  Participants are asked what steps they would take in order to take care of their psychological well-being (for example, spending time with family, or going to a counselor)
Proportion of participants reporting specific motivating/inhibiting factors for taking up therapy | Immediately after treatment (Day 1)
  Participants are asked to select what factors are motivating or inhibiting them in taking up therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- College campus, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data will be posted online

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT06887569/Prot_SAP_000.pdf